CLINICAL TRIAL: NCT06095076
Title: Prospective Descriptive Study of the Cutaneous Microbiota of ICU Patients With Central Venous Catheter (ICMc)
Brief Title: Cutaneous Microbiota Evolution in ICU Patients With CVC (ICMc)
Acronym: ICMc
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Cayenne (Other)
Collaborators: Tropical Biome and ImmunoPhysiopathology (TBIP) - French Guiana University (Université de Guyane) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023_006
Record Dates: First submitted 2023-06-20; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-05

CONDITIONS: Dysbiosis; Catheter-Related Infections
Keywords: Microbiota; Cutaneous microbiota; Healthcare associated infection; Catheter-related infections
MeSH Terms: conditions — Dysbiosis; Catheter-Related Infections; Cross Infection | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skin swab catheter (standard culture)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Skin swabbing — Skin swabbing will be performed on CVC insertion site before CVC placement (baseline), and then every 3 days (or when dressing is changed) while CVC is in place, then at ICU discharge. Bacterial metagenomics using bacterial DNA extraction, 16S PCR amplification and Nanopore sequencing will allow for description of cutaneous microbiota and diversity evaluation through Shannon index. Evolution of alpha-diversity will be evaluated through time-series data analysis: comparison of Shannon index at various time points with baseline Shanonn index (before CVC placement). Standard microbiologic culture of skin swabbing will be performed.
Other: Data collection — General patient characteristics and informations relative to CVC infection and treatment will be collected.

SUMMARY:
Intensive Care Unit (ICU) patients are exposed to catheter-related infections with an important morbidity. Catheter colonization is constant but infection is not. Cutaneous dysbiosis could be the missing link. Our study aims to evaluate the evolution of cutaneous microbiota in ICU patients with a central venous catheter in place, through metagenomics. Our main objective is to evaluate the evolution of alpha-diversity, quantified by intra-patient variation of Shannon diversity index (a diversity index used in bacterial metagenomics).

DETAILED DESCRIPTION:
Central venous catheters (CVCs) are necessary in up to 60% of ICU patients, representing a risk of catheter-related infections with high morbidity and mortality. Catheter colonization originating mostly from the skin is constant, but infection is not. Dysbiosis is known to be associated with pathological states and infection, for example post-antibiotic C. difficile diarrheas, or atopic dermatitis, in which flares are associated with dysbiosis and S. aureus predominance. Cutanous dysbiosis could be the missing link between catheter colonization and infection. Our hypothesis is that under the influence of multiple ICU factors (stress, antibiotic administration, local dysinfection procedures), cutaneous dybiosis appears in ICU patients with a central venous catheter.

All adult ICU patients with an indication for CVC placement will be included over a 6 months period. Skin swabbing will be performed on CVC insertion site before CVC placement (baseline), and then every 3 days (or when dressing is changed) while CVC is in place, then at ICU discharge. Bacterial metagenomics using bacterial DNA extraction, 16S PCR amplification and Nanopore sequencing will allow for description of cutaneous microbiota and diversity evaluation through Shannon index. Evolution of alpha-diversity will be evaluated through time-series data analysis: comparison of Shannon index at various time points with baseline Shanonn index (before CVC placement). Standard microbiologic culture of skin swabbing will be performed. General patient characteristics and informations relative to CVC infection and treatment will be collected.

This study will have no impact on patient management.

Category 3 Non-Interventional Human Person Research (RIPH 3)

ELIGIBILITY:
Inclusion Criteria:

- Adult hospitalized in ICU at the Cayenne Hospital Center in whom the installation of a CVC is indicated

Exclusion Criteria:

* Patient under 18 years of age
* Patient or trusted person or family or relative objecting to participation in the study (refusal)
* Patient under judicial safeguard or under any other protective regime (guardianship or curatorship)
* Patient with cutaneous lesions (infection, burn) near the cutaneous insertion site of the CVC

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult hospitalized in ICU at the Cayenne Hospital Center in whom the installation of a CVC is indicated
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-12-02 (Estimated); Study Completion 2024-06-02 (Estimated)

PRIMARY OUTCOMES:
Evolution of alpha-diversity | Baseline
  Comparison of Shannon index at various time points with baseline Shannon index (before Central Venous Catheter placement through leaving intensive care service). The higher the Shannon index, the greater the diversity.
Evolution of alpha-diversity | Day 3
  Comparison of Shannon index at various time points with baseline Shannon index (before Central Venous Catheter placement through leaving intensive care service). The higher the Shannon index, the greater the diversity.

SECONDARY OUTCOMES:
Skin swabs Metagenomics | Baseline
  Metagenomics: Alpha and beta-diversity of skin swabs
Skin colonization | Baseline
  Skin colonization: positive standard culture of skin swabs
Catheter-related colonization | Baseline
  Catheter-related colonization: standard central line culture positivity
Central Venous Catheter's Metagenomics | Baseline
  Metagenomics: alpha and beta-diversity of Central Venous Catheter at removal
Catheter related Infection | Baseline
  Clinical signs and blood culture and/or positive catheter culture
Skin swabs Metagenomics | Day 3
  Comparison of Shannon index at various time points with baseline Shannon index (before Central Venous Catheter placement through leaving intensive care service). The higher the Shannon index, the greater the diversity.
Skin colonization | Day 3
  Skin colonization: positive standard culture of skin swabs
Catheter-related colonization | Day 3
  Catheter-related colonization: standard central line culture positivity
Central Venous Catheter's Metagenomics | Day 3
  Metagenomics: alpha and beta-diversity of Central Venous Catheter at removal
Catheter related Infection | Day 3
  Clinical signs and blood culture and/or positive catheter culture

CONTACTS AND LOCATIONS:
Overall Officials: Ariane ROUJANSKY, Principal Investigator — Centre Hospitalier de Cayenne
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, Guyane Française, French Guiana

REFERENCES:
- [Background] Tacconelli E, Smith G, Hieke K, Lafuma A, Bastide P. Epidemiology, medical outcomes and costs of catheter-related bloodstream infections in intensive care units of four European countries: literature- and registry-based estimates. J Hosp Infect. 2009 Jun;72(2):97-103. doi: 10.1016/j.jhin.2008.12.012. Epub 2009 Feb 25. PMID 19246122
- [Background] Soufir L, Timsit JF, Mahe C, Carlet J, Regnier B, Chevret S. Attributable morbidity and mortality of catheter-related septicemia in critically ill patients: a matched, risk-adjusted, cohort study. Infect Control Hosp Epidemiol. 1999 Jun;20(6):396-401. doi: 10.1086/501639. PMID 10395140
- [Background] Christensen GD, Simpson WA, Bisno AL, Beachey EH. Adherence of slime-producing strains of Staphylococcus epidermidis to smooth surfaces. Infect Immun. 1982 Jul;37(1):318-26. doi: 10.1128/iai.37.1.318-326.1982. PMID 6179880
- [Background] Safdar N, Maki DG. The pathogenesis of catheter-related bloodstream infection with noncuffed short-term central venous catheters. Intensive Care Med. 2004 Jan;30(1):62-7. doi: 10.1007/s00134-003-2045-z. Epub 2003 Nov 26. PMID 14647886
- [Background] Darouiche RO. Device-associated infections: a macroproblem that starts with microadherence. Clin Infect Dis. 2001 Nov 1;33(9):1567-72. doi: 10.1086/323130. Epub 2001 Sep 26. PMID 11577378
- [Background] Raad I, Costerton W, Sabharwal U, Sacilowski M, Anaissie E, Bodey GP. Ultrastructural analysis of indwelling vascular catheters: a quantitative relationship between luminal colonization and duration of placement. J Infect Dis. 1993 Aug;168(2):400-7. doi: 10.1093/infdis/168.2.400. PMID 8335977
- [Background] Sender R, Fuchs S, Milo R. Revised Estimates for the Number of Human and Bacteria Cells in the Body. PLoS Biol. 2016 Aug 19;14(8):e1002533. doi: 10.1371/journal.pbio.1002533. eCollection 2016 Aug. PMID 27541692
- [Background] Byrd AL, Belkaid Y, Segre JA. The human skin microbiome. Nat Rev Microbiol. 2018 Mar;16(3):143-155. doi: 10.1038/nrmicro.2017.157. Epub 2018 Jan 15. PMID 29332945
- [Background] Coates M, Lee MJ, Norton D, MacLeod AS. The Skin and Intestinal Microbiota and Their Specific Innate Immune Systems. Front Immunol. 2019 Dec 17;10:2950. doi: 10.3389/fimmu.2019.02950. eCollection 2019. PMID 31921196
- [Background] Nakatsuji T, Chen TH, Narala S, Chun KA, Two AM, Yun T, Shafiq F, Kotol PF, Bouslimani A, Melnik AV, Latif H, Kim JN, Lockhart A, Artis K, David G, Taylor P, Streib J, Dorrestein PC, Grier A, Gill SR, Zengler K, Hata TR, Leung DY, Gallo RL. Antimicrobials from human skin commensal bacteria protect against Staphylococcus aureus and are deficient in atopic dermatitis. Sci Transl Med. 2017 Feb 22;9(378):eaah4680. doi: 10.1126/scitranslmed.aah4680. PMID 28228596
- [Background] Grice EA, Kong HH, Conlan S, Deming CB, Davis J, Young AC; NISC Comparative Sequencing Program; Bouffard GG, Blakesley RW, Murray PR, Green ED, Turner ML, Segre JA. Topographical and temporal diversity of the human skin microbiome. Science. 2009 May 29;324(5931):1190-2. doi: 10.1126/science.1171700. PMID 19478181
- [Background] Chen CH, Tu CC, Kuo HY, Zeng RF, Yu CS, Lu HH, Liou ML. Dynamic change of surface microbiota with different environmental cleaning methods between two wards in a hospital. Appl Microbiol Biotechnol. 2017 Jan;101(2):771-781. doi: 10.1007/s00253-016-7846-4. Epub 2016 Oct 22. PMID 27771740
- [Background] Chien AL, Tsai J, Leung S, Mongodin EF, Nelson AM, Kang S, Garza LA. Association of Systemic Antibiotic Treatment of Acne With Skin Microbiota Characteristics. JAMA Dermatol. 2019 Apr 1;155(4):425-434. doi: 10.1001/jamadermatol.2018.5221. PMID 30758497
- [Background] Seekatz AM, Young VB. Clostridium difficile and the microbiota. J Clin Invest. 2014 Oct;124(10):4182-9. doi: 10.1172/JCI72336. Epub 2014 Jul 18. PMID 25036699
- [Background] Kong HH, Oh J, Deming C, Conlan S, Grice EA, Beatson MA, Nomicos E, Polley EC, Komarow HD; NISC Comparative Sequence Program; Murray PR, Turner ML, Segre JA. Temporal shifts in the skin microbiome associated with disease flares and treatment in children with atopic dermatitis. Genome Res. 2012 May;22(5):850-9. doi: 10.1101/gr.131029.111. Epub 2012 Feb 6. PMID 22310478
- [Background] Meylan P, Lang C, Mermoud S, Johannsen A, Norrenberg S, Hohl D, Vial Y, Prod'hom G, Greub G, Kypriotou M, Christen-Zaech S. Skin Colonization by Staphylococcus aureus Precedes the Clinical Diagnosis of Atopic Dermatitis in Infancy. J Invest Dermatol. 2017 Dec;137(12):2497-2504. doi: 10.1016/j.jid.2017.07.834. Epub 2017 Aug 24. PMID 28842320
- [Background] Sommer F, Anderson JM, Bharti R, Raes J, Rosenstiel P. The resilience of the intestinal microbiota influences health and disease. Nat Rev Microbiol. 2017 Oct;15(10):630-638. doi: 10.1038/nrmicro.2017.58. Epub 2017 Jun 19. PMID 28626231
- [Background] Hooks KB, O'Malley MA. Dysbiosis and Its Discontents. mBio. 2017 Oct 10;8(5):e01492-17. doi: 10.1128/mBio.01492-17. PMID 29018121
- [Background] Grice EA, Segre JA. The skin microbiome. Nat Rev Microbiol. 2011 Apr;9(4):244-53. doi: 10.1038/nrmicro2537. PMID 21407241
- [Background] McBride ME, Duncan WC, Knox JM. The environment and the microbial ecology of human skin. Appl Environ Microbiol. 1977 Mar;33(3):603-8. doi: 10.1128/aem.33.3.603-608.1977. PMID 16345214
- [Background] Cusco A, Catozzi C, Vines J, Sanchez A, Francino O. Microbiota profiling with long amplicons using Nanopore sequencing: full-length 16S rRNA gene and the 16S-ITS-23S of the rrn operon. F1000Res. 2018 Nov 6;7:1755. doi: 10.12688/f1000research.16817.2. eCollection 2018. PMID 30815250
- [Background] Haegeman B, Hamelin J, Moriarty J, Neal P, Dushoff J, Weitz JS. Robust estimation of microbial diversity in theory and in practice. ISME J. 2013 Jun;7(6):1092-101. doi: 10.1038/ismej.2013.10. Epub 2013 Feb 14. PMID 23407313
- [Background] Kim BR, Shin J, Guevarra R, Lee JH, Kim DW, Seol KH, Lee JH, Kim HB, Isaacson R. Deciphering Diversity Indices for a Better Understanding of Microbial Communities. J Microbiol Biotechnol. 2017 Dec 28;27(12):2089-2093. doi: 10.4014/jmb.1709.09027. PMID 29032640
- [Background] Timsit JF. [Updating of the 12th consensus conference of the Societe de Reanimation de langue francaise (SRLF): catheter related infections in the intensive care unit]. Ann Fr Anesth Reanim. 2005 Mar;24(3):315-22. doi: 10.1016/j.annfar.2004.12.022. French. PMID 15792575
- [Background] Aagaard K, Petrosino J, Keitel W, Watson M, Katancik J, Garcia N, Patel S, Cutting M, Madden T, Hamilton H, Harris E, Gevers D, Simone G, McInnes P, Versalovic J. The Human Microbiome Project strategy for comprehensive sampling of the human microbiome and why it matters. FASEB J. 2013 Mar;27(3):1012-22. doi: 10.1096/fj.12-220806. Epub 2012 Nov 19. PMID 23165986
- [Background] Rozas M, Brillet F, Callewaert C, Paetzold B. MinION Nanopore Sequencing of Skin Microbiome 16S and 16S-23S rRNA Gene Amplicons. Front Cell Infect Microbiol. 2022 Jan 5;11:806476. doi: 10.3389/fcimb.2021.806476. eCollection 2021. PMID 35071053
- [Background] Matsuo Y, Komiya S, Yasumizu Y, Yasuoka Y, Mizushima K, Takagi T, Kryukov K, Fukuda A, Morimoto Y, Naito Y, Okada H, Bono H, Nakagawa S, Hirota K. Full-length 16S rRNA gene amplicon analysis of human gut microbiota using MinION nanopore sequencing confers species-level resolution. BMC Microbiol. 2021 Jan 26;21(1):35. doi: 10.1186/s12866-021-02094-5. PMID 33499799
- [Background] NCBI Resource Coordinators. Database resources of the National Center for Biotechnology Information. Nucleic Acids Res. 2016 Jan 4;44(D1):D7-19. doi: 10.1093/nar/gkv1290. Epub 2015 Nov 28. PMID 26615191
- [Background] Chen HS, Wang FD, Lin M, Lin YC, Huang LJ, Liu CY. Risk factors for central venous catheter-related infections in general surgery. J Microbiol Immunol Infect. 2006 Jun;39(3):231-6. PMID 16783454
- See also: Santé Publique France- Mission Nationale SPIADI. Surveillance des infections associées aux dispositifs invasifs. Mission nationale SPIADI. Résultats de la surveillance menée en 2019. — https://www.santepubliquefrance.fr/import/surveillance-des-infections-associees-aux-dispositifs-invasifs.-mission-nationale-spiadi.-resultats-de-la-surveillance-menee-en-2019